CLINICAL TRIAL: NCT00337636
Title: A Phase I Study of the Safety and Preliminary Effectiveness of Human CNS Stem Cells (HuCNS-SC) in Patients With Neuronal Ceroid Lipofuscinosis Caused by Palmitoyl Protein Thioesterase 1 (PPT1) or Tripeptidyl Peptidase 1 (TPP-I) Deficiency
Brief Title: Study of HuCNS-SC Cells in Patients With Infantile or Late Infantile Neuronal Ceroid Lipofuscinosis (NCL)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: StemCells, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CL-N001-05
Record Dates: First submitted 2006-06-13; First posted 2006-06-16 (Estimated); Last update posted 2015-01-15 (Estimated); Status verified 2015-01

CONDITIONS: Neuronal Ceroid Lipofuscinosis
Keywords: NCL; INCL; LINCL; Batten disease; Infantile Neuronal Ceroid Lipofuscinosis (INCL); Late Infantile Neuronal Ceroid Lipofuscinosis (LINCL)
MeSH Terms: conditions — Neuronal Ceroid-Lipofuscinoses

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- HuCNS-SC (Experimental): human central nervous system stem cells
  Interventions: Procedure: Surgery to implant human CNS stem cells (HuCNS-SC); Drug: Medication to suppress the immune system

INTERVENTIONS:
Procedure: Surgery to implant human CNS stem cells (HuCNS-SC) — single dose
  Other Names: HuCNS-SC
Drug: Medication to suppress the immune system — Immunosuppression for 12 months post transplant

SUMMARY:
Patients with infantile or late infantile NCL have either a reduced amount of, or are missing, the palmitoyl protein thioesterase 1 (PPT1) enzyme or the tripeptidyl peptidase 1 (TPP-I) enzyme. Human central nervous system stem cells (HuCNS-SC) are an investigational product derived from human brain cells. HuCNS-SC have been shown to survive and migrate within the brains of mice. When grown in the laboratory, HuCNS-SC have been shown to produce the PPT1 and TPP-I enzymes. In mice missing the PPT1 enzyme, HuCNS-SC have been shown to increase the amount of this enzyme in the brain, to reduce the amount of abnormal storage material in the brain, and to prevent the death of some neurons (a type of cell) in the brain.

Participation in this study will involve screening assessments, surgery to implant HuCNS-SC, medication to suppress the immune system, and a series of follow-up assessments. The length of time from the start of screening through to the last follow-up visit will be approximately 13 months, with frequent visits to the study center during this time. After completion of this study, patients will be monitored for an additional 4 years under a separate long term follow-up protocol.

ELIGIBILITY:
Inclusion Criteria:

Patients MAY be eligible to participate in this research study if they:

* Are age 18 months to 12 years old
* Have a clinical diagnosis of infantile neuronal ceroid lipofuscinosis (INCL) or late infantile neuronal ceroid lipofuscinosis (LINCL)
* Have a mutation of the CLN1 or CLN2 gene
* Have severe cognitive, communication, behavior and language impairment

Exclusion Criteria:

Patients may not be eligible to participate in this research study if they:

* Have cognitive, communication, behavior and language function less than that of a 1 year old
* Have previously received an organ, tissue or bone marrow transplantation
* Have previously participated in any gene or cell therapy study
* Have infection with hepatitis virus, Cytomegalovirus, Epstein Barr Virus, or Human Immunodeficiency Virus (HIV)
* Have a current or prior cancer
* Have a bleeding disorder
* Are unable to have an MRI scan

Ages: 18 Months to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 6 (Actual)
Dates: Start 2006-05; Primary Completion 2009-02 (Actual); Study Completion 2009-09 (Actual)

PRIMARY OUTCOMES:
Safety | one year post transpant

SECONDARY OUTCOMES:
Preliminary efficacy | one year post transplant

CONTACTS AND LOCATIONS:
Overall Officials: Robert Steiner, MD, Principal Investigator — Oregon Health and Science University
Locations (1):
- Oregon Health and Science University, Portland, Oregon, United States

REFERENCES:
- [Derived] Selden NR, Al-Uzri A, Huhn SL, Koch TK, Sikora DM, Nguyen-Driver MD, Guillaume DJ, Koh JL, Gultekin SH, Anderson JC, Vogel H, Sutcliffe TL, Jacobs Y, Steiner RD. Central nervous system stem cell transplantation for children with neuronal ceroid lipofuscinosis. J Neurosurg Pediatr. 2013 Jun;11(6):643-52. doi: 10.3171/2013.3.PEDS12397. Epub 2013 Apr 12. PMID 23581634
- See also: Click here for information about StemCells, Inc. — http://www.stemcellsinc.com